CLINICAL TRIAL: NCT06739928
Title: A Safety and Efficacy Evaluation Study of Irinotecan Liposome (II) or Etoposide Combined With Adebrelimab and Carboplatin in the Treatment of ES-SCLC
Brief Title: Irinotecan Liposome (II) or Etoposide Combined With Adebrelimab and Carboplatin in the Treatment of ES-SCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Zhou Chengzhi, doctor, Guangzhou Institute of Respiratory Disease
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES-2024-209-01
Record Dates: First submitted 2024-12-04; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Small Cell Lung Cancer Extensive Stage
Keywords: ES-SCLC; extensive stage-small cell lung cancer; adebrelimab; Irinotecan liposome (II); zhou chengzhi
MeSH Terms: interventions — irinotecan sucrosofate; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irinotecan liposome (II)+adebrelimab+carboplatin (Experimental): The patient received treatment with Irinotecan liposome (II), adebrelimab, and carboplatin.
  Interventions: Drug: Irinotecan liposome (II) combined with adebrelimab and carboplatin
- etoposide+adebrelimab+carboplatin (Other): The patient received treatment with etoposide, adebrelimab, and carboplatin.
  Interventions: Drug: etoposide combined with adebrelimab and carboplatin

INTERVENTIONS:
Drug: Irinotecan liposome (II) combined with adebrelimab and carboplatin — Irinotecan liposome (II) + adebrelimab + carboplatin
  Arms: Irinotecan liposome (II)+adebrelimab+carboplatin
Drug: etoposide combined with adebrelimab and carboplatin — etoposide + adebrelimab + carboplatin
  Arms: etoposide+adebrelimab+carboplatin

SUMMARY:
This study is a prospective, randomized, parallel, multicenter phase II study aimed at evaluating the efficacy and safety of irinotecan liposome (II) or etoposide combined with adebrelimab and carboplatin as first-line treatment for extensive stage small cell lung cancer. The primary endpoint of the study was the 1-year overall survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed small cell lung cancer (SCLC), staged as extensive-stage SCLC (ES-SCLC) according to the VALG staging system;
* No prior systemic treatment received;
* At least a 6-month interval between the last treatment (radiation therapy and chemotherapy) and diagnosis of extensive-stage SCLC;
* Showing at least one target lesion (RECIST 1.1) that has not been previously irradiated;
* Male or female patients aged ≥18 and ≤70 years;
* ECOG performance status (PS) score of 0 or 1;
* Life expectancy of ≥12 weeks;
* Adequate organ function: (1) Hematologic: WBC ≥ 3.0 × 10⁹/L, ANC ≥ 1.5 × 10⁹/L, PLT ≥ 100 × 10⁹/L, HGB ≥ 9.0 g/dL.(2) Hepatic function: AST ≤ 2.5 × ULN, ALT ≤ 2.5 × ULN, liver metastases allowed if ALT and AST ≤ 5 × ULN, TBIL ≤ 1.5 × ULN (except for Gilbert's syndrome, where total bilirubin ≤ 3.0 mg/dL),(3) Renal function: Cr ≤ 1.5 × ULN or CrCl ≥ 50 mL/min, (4) Coagulation: INR ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN;
* Agreement to use an appropriate contraceptive method from the first dose of the study treatment until 6 months after the last dose of the study treatment. Women of childbearing potential must have a negative pregnancy test within 7 days prior to enrollment;
* The patient must have fully understood the study and voluntarily consent to participate by signing the informed consent form (ICF).

Exclusion Criteria:

* Histologically or cytologically confirmed mixed small cell lung cancer (SCLC) and non-small cell lung cancer (NSCLC);
* Previous treatment with immune checkpoint inhibitors, or treatment with irinotecan or other DNA topoisomerase inhibitors;
* Use of a strong CYP3A4 inducer within 2 weeks prior to the first dose of the investigational drug, or a strong CYP3A4 inhibitor or UGT1A1 inhibitor within 1 week prior to the first dose;
* Presence of clinically symptomatic brain metastasis, leptomeningeal metastasis, or spinal cord compression;
* Hematologic disorders, including but not limited to lymphoma, acute or chronic leukemia, multiple myeloma, aplastic anemia, myelodysplastic syndrome, etc;
* Clinically symptomatic third-space fluid accumulation, such as pericardial effusion, pleural effusion, or ascites that cannot be controlled by drainage or other treatments;
* Active, known, or suspected autoimmune disease;
* Use of corticosteroids (doses> 10 mg/day of prednisone or equivalent) or other immunosuppressive agents within 14 days prior to the first dose of the study drug;
* Receipt of live vaccines or planned vaccination with a live vaccine within 4 weeks prior to the first dose of the study drug;
* Interstitial lung disease, drug-induced pneumonia, radiation-induced pneumonia requiring steroid treatment, or clinically symptomatic active pneumonia, or severe pulmonary dysfunction;
* Active tuberculosis or a history of active tuberculosis within 48 weeks prior to screening, regardless of whether it was treated;
* Any toxicity from previous anticancer therapy, that has not resolved to grade ≤1 (according to CTCAE v5.0) prior to the first dose of the investigational drug;
* Underwent a minor surgery (including catheter placement) within 48 hours prior to the first dose of the study drug;
* Presence of uncontrolled cardiovascular symptoms or diseases;
* Hypersensitivity to the investigational drug or its excipients;
* A history of any other malignancy within 5 years prior to the first dose of the study drug, except for adequately treated non-melanoma skin cancer or in situ carcinoma;
* A history of psychiatric disorders, alcohol abuse, drug abuse, or substance misuse;
* HBsAg-positive and HBV DNA levels exceeding the upper limit of normal, or HCV-positive (HCV RNA or HCV Ab indicating acute or chronic infection); a history of HIV-positive status or acquired immunodeficiency syndrome (AIDS);
* Received any other investigational drug or participated in another interventional clinical trial within 4 weeks prior to signing the informed consent form (ICF);
* A history of allogeneic bone marrow transplantation or solid organ transplantation;
* Any other factors as determined by the investigator.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
1-year OS rate | 1 year
  The proportion of patients who are still alive after one year of treatment.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 1 year
  Time from start of patient's treatment to disease progression or death from any cause.
Overall survival (OS) | 2 years
  Time from patient randomization to patient death from any cause.
Objective response rate (ORR) | 1 year
  Proportion of patients whose tumor volume shrinks to a pre-specified value and who can maintain the minimum timeframe requirement, as the sum of the proportion in complete and partial remission.
Disease control rate（DCR） | 1 year
  Number of cases in remission (PR+CR) and stable lesions (SD) after treatment as a percentage of evaluable cases.
Duration of Response (DoR) | 1 year
  the time between the first time a subject in confirmed complete remission (CR) or confirmed partial remission (PR) reaches confirmed complete remission (CR) or confirmed partial remission (PR) and the time of the first disease progression or death of any cause.
AEs rate | 3 years.
  Incidence of adverse events occurring during treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Chengzhi Zhou, Doctor, Principal Investigator — Guangzhou Institute of Respiratory Disease (Responsible Party)
Locations (1):
- Guangzhou Institute of Respiratory Disease (Responsible Party), Guangzhou, Guangzhou, China